CLINICAL TRIAL: NCT07028164
Title: Epidemiology, Prognosis, and Treatment Effectiveness of Asymptomatic Biliary Dilatation
Brief Title: Clinical Features and Prognosis of Asymptomatic Biliary Dilatation
Status: Completed | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Shuo Jin, Associate Chief Physician, Beijing Tsinghua Chang Gung Hospital
Other Study IDs: 24640-0-01-1
Record Dates: First submitted 2025-06-02; First posted 2025-06-19 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Choledochal Cyst
Keywords: Cohort study; Clinical database; Surgical treatment; Long-term outcome; Asymptomatic Biliary Dilatation; Natural outcome
MeSH Terms: conditions — Choledochal Cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: This cohort retrospectively collects all available clinical data and prognostic information of all patients who were previously diagnosed with asymptomatic biliary dilatation in the participating centers, and compares the various outcome indicators of two groups or multiple groups.
- Prospective cohort: This cohort prospectively enrolls all patients with a clear diagnosis of biliary dilatation in each participating center, tracks and observes them for a certain period of time, and compares the various outcome indicators of two groups or multiple groups. Additionally, it conducts prospective follow-ups on the patients in the retrospective cohort.

SUMMARY:
This study is a multicenter, ambidirectional cohort study aiming to consecutively recruit asymptomatic biliary dilation patients incidentally discovered by imaging from 25 medical centers across China. The investigators will collect comprehensive clinicopathological data from the cohort to evaluate the epidemiological characteristics of asymptomatic patients, the distribution of Todani classifications, common imaging-detected comorbidities, and natural history; and, based on high-quality evidence, assess whether surgical intervention can improve the prognosis of asymptomatic patients, thereby providing a basis for developing targeted surveillance and intervention strategies.

DETAILED DESCRIPTION:
Biliary dilation (BD) is a common and complex benign biliary disorder, for which surgical resection remains the only definitive treatment. However, while there are numerous studies on symptomatic BD, there is a lack of systematic, reliable data that describing the population structure, complication rates, comparing natural history and postoperative outcomes of patients whom incidentally detected by imaging and have no biliary symptoms. This multicenter, ambidirectional cohort study aims to consecutively recruit asymptomatic BD patients from 25 tertiary medical centers across China and to systematically collect their clinicopathological data-including demographic characteristics, baseline clinical features, laboratory and imaging results, biliary specific biomarkers, and longitudinal follow up records-in order to establish an asymptomatic subcohort within the larger China BD cohort. Based on this subcohort, the research objectives are structured as follows:

1. Database Establishment and Maintenance: Construct and continuously update a multicenter clinical database for asymptomatic BD patients in China, ensuring data completeness and accessibility.
2. Epidemiological Characterization of Asymptomatic BD: Describe the epidemiological features of asymptomatic BD patients, including demographic profiles (age, sex), distribution of Todani classifications, incidence of various complications, and risk of malignant transformation.
3. Comparison of Surgical Treatment Versus Conservative Observation: Compare key clinical outcomes between asymptomatic BD patients who undergo surgical intervention and those managed by medical observation, thereby providing evidence-based guidance for clinical decision making in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been definitive diagnosed with biliary dilation.
2. Patients aged between 0 and 80 years old, regardless of gender.
3. In line with the principle of informed consent: For the retrospective cohort of biliary dilation, exemption from signing the informed consent form is applied for, while for the prospective cohort, signing the informed consent form is required.

Exclusion Criteria:

-

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a definitive diagnosis of biliary dilation in the participating centers will be included.
Sampling Method: Non-Probability Sample
Enrollment: 1008 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Complications rate | Through study completion, an average of 5 years
  The occurrences of long-term postoperative complications include recurrent cholangitis, pancreatitis, bile duct stones, liver failure, and other such conditions.

SECONDARY OUTCOMES:
Malignant transformation rate | Through study completion, an average of 5 year
  The occurrence of malignant transformation associated with bile duct dilatation.

OTHER OUTCOMES:
Mayo Score | Through study completion, an average of 5 year
  The scoring results are categorized into four levels:
  Excellent: Biochemical tests are normal, no clinical symptoms, no anatomical abnormalities; Good: No signs of cholangitis, only minor biliary structural abnormalities; biochemical indices are normal or near normal; no clinical intervention required; Fair: Mild structural biliary abnormalities; cholangitis episodes occur less than 3 times per year and respond to conservative management (e.g., antibiotics); Poor: Recurrent cholangitis (≥ 3 episodes per year); biliary anatomical anomalies (strictures and stones) not amenable to conservative management, requiring reoperation.
the Patient-Reported Outcomes Measurement Information System (PROMIS-29) Score | Through study completion, an average of 5 year
  Patient-reported quality of life will be assessed using the PROMIS-29 Profile v2.1. This validated instrument consists of 29 items covering seven domains: physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, and pain interference (4 items per domain), as well as one item measuring pain intensity (0-10 numeric rating scale). Each domain score is converted to a standardized T-score (mean = 50, standard deviation = 10) based on general population. Higher scores indicate worse symptoms for anxiety, depression, fatigue, sleep disturbance, and pain interference. Higher scores indicate better status for physical function and social role participation.

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Jin, PhD, Principal Investigator — Beijing Tsinghua Chang Gung Hospital
Locations (1):
- Beijing Tsinghua Chang Gung Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No